CLINICAL TRIAL: NCT01278199
Title: A Multicentric Randomized Trial Comparing the Bronchial Artery Embolization Combined With Medical Measures and the Medical Measures Alone in the Treatment of Non-severe Acute Hemoptysis of Mild-to-moderate Abundance
Brief Title: Bronchial Artery Embolization and Medical Measures in Non Severe Acute Hemoptysis of Mild-moderate Abundance
Acronym: ARTEMHYS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K081202
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Hemoptysis; Acute Disease
Keywords: Bronchial Artery Embolization; Non-severe Hemoptysis; Bleeding mild-to-moderate abundance; Volume ranging from 100 ml to 200 ml
MeSH Terms: conditions — Hemoptysis; Acute Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): Medicals measures in the treatment of non-severe acute hemoptysis
  Interventions: Other: Medicals measures
- 1 (Experimental): bronchial artery embolization (BAE)
  Interventions: Other: bronchial artery embolization

INTERVENTIONS:
Other: Medicals measures — Rest in bed. Monitoring of respiratory frequency. Fixation of intravenous route. Administration of nasal oxygenotherapy in order to maintain SpO2 > 90%. Administration of antituberculosis treatment, in case with active pulmonary tuberculosis known at admission or diagnosed during the stay.
  If necessary a bronchial wash out of will be realized by a bronchial fibroscopy with measures of use of cold serum, adrenalin xylocain or terlipressin.
  The administration of antibiotherapy by general mode according to the clinician appreciation.
  The administration of terlipressin according to the clinician appreciation. Against the cough treatment administration according to the clinician appreciation.
  Arms: 2
Other: bronchial artery embolization — The bronchial artery embolization is practised within 48 hours which follow the hospital admission for non-severe acute hemoptysis.
  Arms: 1

SUMMARY:
Severe hemoptysis is a life-threatening condition, with an unpredictable course. The efficacy of bronchial artery embolization (BAE) is well established for the treatment of severe hemoptysis, with short and long-term bleeding controls obtained in 70 to 100% and 50 to 90% of cases, respectively. As complications related to vascular interventional radiology may occur in 5 to 10% of cases, the benefit-risk balance might be less clear in acute hemoptysis of mild-to-moderate abundance (volume between 100 and 200 ml) and no criteria of severity (respiratory failure or hemodynamic instability). There is no available data comparing the safety and efficacy of BAE combined with medical measures to those of medical measures alone in the treatment of non-severe acute hemoptysis of mild-to-moderate abundance.

DETAILED DESCRIPTION:
The study is a multicentric (n=8) randomized study, involving two parallel groups of patients with non-severe acute hemoptysis of mild-to-moderate abundance, related to a systemic bronchial or non-bronchial hypervascularization, and comparing the bronchial artery embolization combined with medical measures and the medical measures alone in this field.

The primary aim of the study is to evaluate the efficacy of BAE combined with medical measures in the treatment of non-severe acute hemoptysis of mild-to-moderate abundance, as compared with that of medical measures alone, by assessing the percentage of recurrence of hemoptysis at one month. Bleeding recurrence is defined as a volume of blood expectorated of at least 50 ml.

The second objectives of the study are to compare the efficacy of the two strategies at 3 months and to assess the safety of both strategies during hospitalization and follow-up.

Based on a previous study of our group (Reference 8), the number of patients in each group is 105, assuming a one-month bleeding recurrence rate of 11% in the group receiving BAE, as compared with 26% in the group assisted medically (a=.05; β=0.8).

ELIGIBILITY:
Inclusion Criteria:

* Non-severe acute hemoptysis (mild-to-moderate abundance and no criteria of severity).
* Age > 18 years
* Patients with social insurance

Exclusion Criteria:

* Pregnant and/or lactating women
* Traumatic hemoptysis
* Severe hemoptysis (volume > 200 ml; respiratory failure; hemodynamic instability)
* Patients already enrolled in the study within the preceding 3 months
* Patients in palliative care, for whom there is no therapeutic plan at short-term
* Moribund patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-12-27 (Actual); Study Completion 2017-02-27 (Actual)

PRIMARY OUTCOMES:
Bleeding recurrence rate, after initial therapeutic strategy. | One month
  Bleeding recurrence is defined as a volume of expectorated blood of 50 ml or more.

SECONDARY OUTCOMES:
Evaluation of the rate of serious adverse events | 3 months
  Evaluation of the rate of serious adverse events, according to the therapeutic strategy during hospitalization and follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Muriel FARTOUKH, MD, Principal Investigator — Tenon Hospital, AP-HP
Locations (1):
- Tenon Hospital, AP-HP, Paris, France

REFERENCES:
- [Background] Mal H, Rullon I, Mellot F, Brugiere O, Sleiman C, Menu Y, Fournier M. Immediate and long-term results of bronchial artery embolization for life-threatening hemoptysis. Chest. 1999 Apr;115(4):996-1001. doi: 10.1378/chest.115.4.996. PMID 10208199
- [Background] PURSEL SE, LINDSKOG GE. Hemoptysis. A clinical evaluation of 105 patients examined consecutively on a thoracic surgical service. Am Rev Respir Dis. 1961 Sep;84:329-36. doi: 10.1164/arrd.1961.84.3.329. No abstract available. PMID 13738524
- [Background] Hirshberg B, Biran I, Glazer M, Kramer MR. Hemoptysis: etiology, evaluation, and outcome in a tertiary referral hospital. Chest. 1997 Aug;112(2):440-4. doi: 10.1378/chest.112.2.440. PMID 9266882
- [Background] Revel MP, Fournier LS, Hennebicque AS, Cuenod CA, Meyer G, Reynaud P, Frija G. Can CT replace bronchoscopy in the detection of the site and cause of bleeding in patients with large or massive hemoptysis? AJR Am J Roentgenol. 2002 Nov;179(5):1217-24. doi: 10.2214/ajr.179.5.1791217. PMID 12388502
- [Background] Mal H. [Role of surgery in the management of severe haemoptysis]. Rev Mal Respir. 2005 Nov;22(5 Pt 1):717-9. doi: 10.1016/s0761-8425(05)85627-x. No abstract available. French. PMID 16272972
- [Background] Picard C, Parrot A, Boussaud V, Lavole A, Saidi F, Mayaud C, Carette MF. Massive hemoptysis due to Rasmussen aneurysm: detection with helicoidal CT angiography and successful steel coil embolization. Intensive Care Med. 2003 Oct;29(10):1837-9. doi: 10.1007/s00134-003-1912-y. Epub 2003 Sep 13. PMID 13680121
- [Background] Remy J, Lemaitre L, Lafitte JJ, Vilain MO, Saint Michel J, Steenhouwer F. Massive hemoptysis of pulmonary arterial origin: diagnosis and treatment. AJR Am J Roentgenol. 1984 Nov;143(5):963-9. doi: 10.2214/ajr.143.5.963. PMID 6333165
- [Background] Fartoukh M, Khalil A, Louis L, Carette MF, Bazelly B, Cadranel J, Mayaud C, Parrot A. An integrated approach to diagnosis and management of severe haemoptysis in patients admitted to the intensive care unit: a case series from a referral centre. Respir Res. 2007 Feb 15;8(1):11. doi: 10.1186/1465-9921-8-11. PMID 17302979
- [Background] Savale L, Parrot A, Khalil A, Antoine M, Theodore J, Carette MF, Mayaud C, Fartoukh M. Cryptogenic hemoptysis: from a benign to a life-threatening pathologic vascular condition. Am J Respir Crit Care Med. 2007 Jun 1;175(11):1181-5. doi: 10.1164/rccm.200609-1362OC. Epub 2007 Mar 1. PMID 17332480
- [Background] Bruzzi JF, Remy-Jardin M, Delhaye D, Teisseire A, Khalil C, Remy J. Multi-detector row CT of hemoptysis. Radiographics. 2006 Jan-Feb;26(1):3-22. doi: 10.1148/rg.261045726. PMID 16418239
- [Background] Khalil A, Parrot A, Nedelcu C, Fartoukh M, Marsault C, Carette MF. Severe hemoptysis of pulmonary arterial origin: signs and role of multidetector row CT angiography. Chest. 2008 Jan;133(1):212-9. doi: 10.1378/chest.07-1159. Epub 2007 Nov 7. PMID 17989162
- [Background] Dweik RA, Stoller JK. Role of bronchoscopy in massive hemoptysis. Clin Chest Med. 1999 Mar;20(1):89-105. doi: 10.1016/s0272-5231(05)70129-5. PMID 10205720
- [Background] Crocco JA, Rooney JJ, Fankushen DS, DiBenedetto RJ, Lyons HA. Massive hemoptysis. Arch Intern Med. 1968 Jun;121(6):495-8. No abstract available. PMID 5652400
- [Background] Garzon AA, Cerruti MM, Golding ME. Exsanguinating hemoptysis. J Thorac Cardiovasc Surg. 1982 Dec;84(6):829-33. PMID 7144217
- [Background] Jewkes J, Kay PH, Paneth M, Citron KM. Pulmonary aspergilloma: analysis of prognosis in relation to haemoptysis and survey of treatment. Thorax. 1983 Aug;38(8):572-8. doi: 10.1136/thx.38.8.572. PMID 6612647
- [Background] Knott-Craig CJ, Oostuizen JG, Rossouw G, Joubert JR, Barnard PM. Management and prognosis of massive hemoptysis. Recent experience with 120 patients. J Thorac Cardiovasc Surg. 1993 Mar;105(3):394-7. PMID 8445918
- [Background] Hakanson E, Konstantinov IE, Fransson SG, Svedjeholm R. Management of life-threatening haemoptysis. Br J Anaesth. 2002 Feb;88(2):291-5. doi: 10.1093/bja/88.2.291. PMID 11878664
- [Background] Jean-Baptiste E. Clinical assessment and management of massive hemoptysis. Crit Care Med. 2000 May;28(5):1642-7. doi: 10.1097/00003246-200005000-00066. PMID 10834728
- [Background] Lordan JL, Gascoigne A, Corris PA. The pulmonary physician in critical care * Illustrative case 7: Assessment and management of massive haemoptysis. Thorax. 2003 Sep;58(9):814-9. doi: 10.1136/thorax.58.9.814. No abstract available. PMID 12947147
- [Background] Haponik EF, Chin R. Hemoptysis: clinicians' perspectives. Chest. 1990 Feb;97(2):469-75. doi: 10.1378/chest.97.2.469. PMID 2298074
- [Background] Haponik EF, Fein A, Chin R. Managing life-threatening hemoptysis: has anything really changed? Chest. 2000 Nov;118(5):1431-5. doi: 10.1378/chest.118.5.1431. PMID 11083697
- [Background] Remy J, Arnaud A, Fardou H, Giraud R, Voisin C. Treatment of hemoptysis by embolization of bronchial arteries. Radiology. 1977 Jan;122(1):33-7. doi: 10.1148/122.1.33. PMID 830351
- [Background] Ramon P, Wallaert B, Derollez M, D'Odemont JP, Tonnel AB. [Treatment of severe hemoptysis with terlipressin. Study of the efficacy and tolerance of this product]. Rev Mal Respir. 1989;6(4):365-8. French. PMID 2799045
- [Background] White RI Jr. Bronchial artery embolotherapy for control of acute hemoptysis: analysis of outcome. Chest. 1999 Apr;115(4):912-5. doi: 10.1378/chest.115.4.912. No abstract available. PMID 10208183
- [Background] Remy J, Voisin C, Dupuis C, Beguery P, Tonnel AB, Denies JL, Douay B. [Treatment of hemoptysis by embolization of the systemic circulation]. Ann Radiol (Paris). 1974 Jan-Feb;17(1):5-16. No abstract available. French. PMID 4820232
- [Background] Cremaschi P, Nascimbene C, Vitulo P, Catanese C, Rota L, Barazzoni GC, Cornalba GP. Therapeutic embolization of bronchial artery: a successful treatment in 209 cases of relapse hemoptysis. Angiology. 1993 Apr;44(4):295-9. doi: 10.1177/000331979304400405. PMID 8457080
- [Background] Uflacker R, Kaemmerer A, Picon PD, Rizzon CF, Neves CM, Oliveira ES, Oliveira ME, Azevedo SN, Ossanai R. Bronchial artery embolization in the management of hemoptysis: technical aspects and long-term results. Radiology. 1985 Dec;157(3):637-44. doi: 10.1148/radiology.157.3.4059552.
- [Background] Mesurolle B, Lacombe P, Barre O, Qanadli S, Mulot RO, Chagnon S. [Failures and complications of bronchial artery embolization]. Rev Mal Respir. 1996 Jul;13(3):217-25. French. PMID 8765913
- [Background] Ramakantan R, Bandekar VG, Gandhi MS, Aulakh BG, Deshmukh HL. Massive hemoptysis due to pulmonary tuberculosis: control with bronchial artery embolization. Radiology. 1996 Sep;200(3):691-4. doi: 10.1148/radiology.200.3.8756916.
- [Background] Rabkin JE, Astafjev VI, Gothman LN, Grigorjev YG. Transcatheter embolization in the management of pulmonary hemorrhage. Radiology. 1987 May;163(2):361-5. doi: 10.1148/radiology.163.2.3562815.
- [Background] Hayakawa K, Tanaka F, Torizuka T, Mitsumori M, Okuno Y, Matsui A, Satoh Y, Fujiwara K, Misaki T. Bronchial artery embolization for hemoptysis: immediate and long-term results. Cardiovasc Intervent Radiol. 1992 May-Jun;15(3):154-8; discussion 158-9. doi: 10.1007/BF02735578. PMID 1628281
- [Background] Swanson KL, Johnson CM, Prakash UB, McKusick MA, Andrews JC, Stanson AW. Bronchial artery embolization : experience with 54 patients. Chest. 2002 Mar;121(3):789-95. doi: 10.1378/chest.121.3.789. PMID 11888961
- [Background] Wong ML, Szkup P, Hopley MJ. Percutaneous embolotherapy for life-threatening hemoptysis. Chest. 2002 Jan;121(1):95-102. doi: 10.1378/chest.121.1.95. PMID 11796437
- [Background] Ong TH, Eng P. Massive hemoptysis requiring intensive care. Intensive Care Med. 2003 Feb;29(2):317-20. doi: 10.1007/s00134-002-1553-6. Epub 2002 Nov 2. PMID 12594593
- [Background] Labbe V, Roques S, Boughdene F, Razazi K, Khalil A, Parrot A, Fartoukh M. Shock complicating successful bronchial artery embolization for severe hemoptysis. Chest. 2009 Jan;135(1):215-217. doi: 10.1378/chest.08-0491. PMID 19136409
- [Background] Lacerda JE, Consolim-Colombo FM, Moreira ED, Ida F, Silva GJ, Irigoyen MC, Krieger EM. Influence of cardiopulmonary reflex on the sympathetic activity during myocardial infarction. Auton Neurosci. 2007 May 30;133(2):128-35. doi: 10.1016/j.autneu.2006.10.009. Epub 2006 Dec 26. PMID 17188942
- [Background] Remy-Jardin M, Bouaziz N, Dumont P, Brillet PY, Bruzzi J, Remy J. Bronchial and nonbronchial systemic arteries at multi-detector row CT angiography: comparison with conventional angiography. Radiology. 2004 Dec;233(3):741-9. doi: 10.1148/radiol.2333040031. Epub 2004 Oct 14. PMID 15486218
- [Background] Yoon YC, Lee KS, Jeong YJ, Shin SW, Chung MJ, Kwon OJ. Hemoptysis: bronchial and nonbronchial systemic arteries at 16-detector row CT. Radiology. 2005 Jan;234(1):292-8. doi: 10.1148/radiol.2341032079. Epub 2004 Nov 18. PMID 15550375
- [Background] Straus DJ, Yahalom J, Gaynor J, Myers J, Koziner B, Caravelli J, Lee BJ 3rd, Nisce LZ, McCormick B, Bajorunas D, et al. Four cycles of chemotherapy and regional radiation therapy for clinical early-stage and intermediate-stage Hodgkin's disease. Cancer. 1992 Feb 15;69(4):1052-60. doi: 10.1002/1097-0142(19920215)69:43.0.co;2-9. PMID 1370915
- [Background] JACKSON GG, ARANA-SIALER JA, ANDERSEN BR GRIEBLE HG, McCABE WR. Profiles of pyelonephritis. Arch Intern Med. 1962 Nov;110:63-75. No abstract available. PMID 13957202
- [Derived] Fartoukh M, Demoule A, Sanchez O, Tuffet S, Bergot E, Godet C, Andrejak C, Pontier-Marchandise S, Parrot A, Mayaux J, Meyer G, Cluzel P, Sapoval M, Le Pennec V, Carette MF, Cadranel J, Rousseau A, Khalil A, Simon T; ARTEMHYS trial group. Randomised trial of first-line bronchial artery embolisation for non-severe haemoptysis of mild abundance. BMJ Open Respir Res. 2021 Jun;8(1):e000949. doi: 10.1136/bmjresp-2021-000949. PMID 34088727